CLINICAL TRIAL: NCT02893605
Title: Study of Gene Polymorphisms Involved in the Metabolism and Action of Vitamin D in Amyotrophic Lateral Sclerosis
Acronym: SLA_Vit_D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2014/KM-01
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients have a sporadic form of Amyotrophic Lateral Sclerosis.
- Controls: Controls correspond to spouses/partners of patients.

SUMMARY:
This is a case-control study performed on a biological collection. The polymorphisms present on a pre-defined list of genes will be studied for 400 Amyotrophic Lateral Sclerosis (sporadic type) DNA samples and 400 control DNA samples.

ELIGIBILITY:
Inclusion Criteria:

* The primary inclusion criterium is the same for that of the parent biological collection, i.e. the patients fulfill requirements for probable or definite Amyotrophic Lateral Sclerosis as defined by revised international criteria (Brooks et al 2000).
* Additionally, included patients were followed-up by doctors at the University Hospital of Montpellier, thus enabling verification of Amyotrophic Lateral Sclerosis criteria over time.

Exclusion Criteria:

* The patient has a familial form of Amyotrophic Lateral Sclerosis (autosomic dominant or recessive types) with or without a mutation of one of the 3 genes known to be responsible for familial forms (SOD1, TARDBP, FUS). See Bender (1998).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A national biological (France) collection has been in existence since 1996 and serves as a source for patient and control samples. Patients have a sporadic form of Amyotrophic Lateral Sclerosis and controls are their spouses/partners.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-03; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The polymorphisms occurring on a pre-defined set of genes | Day 0 (transversal study)
  The genes studied are: CYP2R1, CYP27A1, CYP3A4, CYP2J2, CYP27B1, CYP24A1, VDBP, VDR.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mouzat, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier, France

REFERENCES:
- [Result] Mouzat K, Raoul C, Polge A, Kantar J, Camu W, Lumbroso S. Liver X receptors: from cholesterol regulation to neuroprotection-a new barrier against neurodegeneration in amyotrophic lateral sclerosis? Cell Mol Life Sci. 2016 Oct;73(20):3801-8. doi: 10.1007/s00018-016-2330-y. Epub 2016 Aug 10. PMID 27510420